CLINICAL TRIAL: NCT03820336
Title: Cardiovascular Effects of Extra Virgin Olive Oil (EVOO) in Healthy Reproductive-aged Women: A Randomized Controlled Trial
Brief Title: Cardiovascular Effects of EVOO in Healthy Reproductive-aged Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Erin Morris, Assistant Professor, Maternal-Fetal Medicine, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18-0639
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hypertension; Vascular Stiffness
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra Virgin Olive Oil (Experimental)
  Interventions: Dietary Supplement: Extra Virgin Olive Oil
- Control Oil (Placebo Comparator)
  Interventions: Dietary Supplement: Control Oil

INTERVENTIONS:
Dietary Supplement: Extra Virgin Olive Oil — Subjects will consume 45 ml (40 g) of EVOO daily for 8 weeks.
  Arms: Extra Virgin Olive Oil
Dietary Supplement: Control Oil — Subjects will consume 45 ml (40 g) of a control sunflower seed oil daily for 8 weeks.
  Arms: Control Oil

SUMMARY:
This study aims to compare changes in cardiovascular function and markers of inflammation and metabolic dysfunction in women randomized to treatment with extra virgin olive oil (EVOO) versus those randomized to treatment with a control oil low in oleic acid and phenols for 8 weeks.

DETAILED DESCRIPTION:
Participants will be randomized to receive 45 ml (40 g) of extra virgin olive oil (EVOO) daily for 8 weeks or an identical dose of a control sunflower seed oil low in oleic acid and phenol content. EVOO high in oleic acid and phenolic content will be identified and shipped from Italy and stored protected from heat and light in the Bionutrition Core at the Clinical Research Center at the University of Vermont Medical Center. Women will undergo a detailed cardiovascular assessment at baseline and following treatment, including assessment of blood pressure, pulse-wave velocity, calculation of arterial distensibility and beta stiffness, flow-mediated vasodilation, cardiac output, response to volume challenge and dual-energy X-ray absorptiometry (DEXA). Lipid profiles and markers of inflammation, oxidative stress and metabolic dysfunction will also be assessed at both study visits.

Investigators hypothesize that treatment with high oleic acid and phenolic EVOO will be associated with decreased blood pressure, improved vascular compliance and blood vessel function, and with improvement in lipid profile, inflammation and markers of metabolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Women are eligible to participate if they are between the ages of 18 and 40, in good health, with regular menstrual cycles and no prior pregnancies.

Exclusion Criteria:

* Routinely take medications or supplements known to affect blood pressure, heart or blood vessel function, or those with anti-inflammatory or antioxidant properties
* Smoking
* Pregnancy
* Other conditions that would impair adherence, such as allergy to olive oil or sunflower oil or difficulty swallowing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Arterial pulse wave velocity | 8 weeks
  Arterial pulse wave velocity in meters/second. This is an index of vessel stiffness.
Blood pressure | 8 weeks
  Blood pressure in millimeters mercury (mm Hg).
Arterial distensibility | 8 weeks
  Arterial distensibility (no units). This is an index of vessel stiffness.
Arterial Beta Stiffness Index | 8 weeks
  Arterial Beta Stiffness Index (no units). This is an index of vessel stiffness.

SECONDARY OUTCOMES:
Flow-mediated vasodilation | 8 weeks
  Flow-mediated vasodilation in percent. This is a measure of endothelial health.
Cardiac output | 8 weeks
  Cardiac output in liters per minute.
Cardiac output response to volume challenge | 8 weeks
  Cardiac output response to volume challenge in liters per minute. This is a measure of vascular compliance.
C-reactive protein | 1 year
  Serum C-reactive protein in milligrams/liter. This is a marker of inflammation.
High Density Lipoprotein (HDL) Cholesterol | 1 year
  Serum high density lipoprotein in milligrams/deciliter.
Low Density Lipoprotein (LDL) Cholesterol | 1 year
  Serum low density lipoprotein in milligrams/deciliter.
Triglycerides | 1 year
  Serum triglycerides in milligrams/deciliter.
Insulin | 1 year
  Fasting serum insulin level in micro international units per milliliter (µIU/mL).
Hemoglobin A1C | 1 year
  Serum hemoglobin A1C in percent.
B-type natriuretic peptide (BNP) | 1 year
  B-type natriuretic peptide (BNP) in picograms per milliliter. This is a measure of cardiac function.
Interleukin 6 (IL-6) | 1 year
  Interleukin 6 in picograms per milliliter. This is a measure of inflammation.
Tumor necrosis factor alpha (TNF-α) | 1 year
  Tumor necrosis factor alpha in picograms per milliliter. This is a measure of inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Erin A Morris, MD, Principal Investigator — University of Vermont Medical Center
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No